CLINICAL TRIAL: NCT02924467
Title: Centralized IIS-based Reminder/Recall to Increase Childhood Influenza Vaccination Rates in New York State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-001552; 1R01AI114903 (NIH)
Record Dates: First submitted 2016-09-23; First posted 2016-10-05 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Reminder System for Influenza Vaccines
Keywords: reminder systems; Influenza vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- No intervention: Usual Care (No Intervention): Patients in this group will not receive any influenza vaccine reminder notifications.
- 1 Notice (Experimental): Patients in this group will receive one influenza vaccine reminder notification via autodialer across the 2016 influenza season.
  Interventions: Behavioral: 1 Notice
- 2 Notices (Experimental): Patients in this group will receive up to two influenza vaccine reminder notifications via autodialer throughout the 2016 influenza season.
  Interventions: Behavioral: 2 Notices
- 3 Notices (Experimental): Patients in this group will receive up to three influenza vaccine reminder notifications via autodialer throughout the 2016 influenza season.
  Interventions: Behavioral: 3 Notices

INTERVENTIONS:
Behavioral: 1 Notice — 1 Reminder notification via autodialer
  Other Names: reminders, notifications
  Arms: 1 Notice
Behavioral: 2 Notices — 2 Reminder notifications via autodialer
  Arms: 2 Notices
Behavioral: 3 Notices — 3 Reminder notifications via autodialer
  Arms: 3 Notices

SUMMARY:
Despite U.S. guidelines for influenza vaccination of all children starting at age 6 months, only about half of children are vaccinated annually, leading to substantial influenza disease in children and spread of disease to adults. A major barrier is that families are not reminded about the need for their children to receive influenza vaccination. The investigators will evaluate the impact of patient reminder/recall performed by state immunization information systems to improve influenza vaccination rates by using three clinical trials in two states. The investigators will assess effectiveness and cost-effectiveness of phone reminder/recall on improving influenza vaccination rates. The investigators will disseminate the state immunization information system-based reminder/recall system to all states for use for seasonal and pandemic influenza vaccinations with the goal of lowering influenza morbidity.

DETAILED DESCRIPTION:
Annual epidemics of influenza A and B cause substantial morbidity and mortality in the US with high rates of hospitalizations, emergency department visits, outpatient visits, and medical costs. Children experience significant morbidity from influenza and also play a key role in instigating and expanding epidemics. In addition, concerns about pandemic influenza heighten the importance of new mechanisms to rapidly inform the population about influenza and direct efforts for rapid vaccine delivery.

Since 2010, the Advisory Committee on Immunization Practices (ACIP) has recommended influenza vaccination for all children >6 months of age. However, vaccination rates remain very low. For the 2012-2013 season, only 56% of children 2-17y were vaccinated. Modeling studies suggest that as many as 19 million cases of influenza could be prevented if child vaccination rates were raised to 70% nationally. The most effective strategy recommended by CDC and the Task Force on Community Preventive Services for improving childhood influenza vaccination rates is reminder/recall (R/R), sent by phone or mail, notifying parents of the need to vaccinate their child. The published literature suggests R/R can improve influenza vaccination rates. However, few practices use R/R; barriers are practice costs, insufficient staff time and expertise, and lack of predictability regarding receipt of vaccine supplies.

Statewide immunization information systems (IISs) now exist in all states to track vaccinations. They have not yet been used for influenza vaccine R/R because of lack of evidence for their effectiveness and a lack of a template for IIS-based reminder/recall. The investigators have united two leading immunization research groups (Denver, CO and Rochester, NY) to assess the impact of centralized IIS-based influenza vaccine reminder/recall, and to evaluate the effect of intensity of recall (1 v. 2. v. 3 reminders) over usual care. The investigators will also develop tools to aid other states in creating efficient IIS reminder/recall systems. The investigators will also develop tools to aid other states in creating efficient IIS reminder/recall systems for seasonal and possible pandemic influenza outbreaks.

The study has four aims:

Aim 1 is to develop the protocols, clinical decision support, and message content for state IISs to conduct reminder/recall for influenza vaccinations.

Aim 2 is to conduct a pragmatic trial, with randomization at the level of the patient within practices randomly selected to be proportionate to each state, to compare: 1) effectiveness and cost-effectiveness of centralized reminder/recall of different intensity (1 v.2 v. 3 messages) and usual care (0 messages) and 2) effectiveness and cost-effectiveness of reminder/recall in specified subgroups (family medicine vs. pediatric provider, rural vs urban, age of child) on receipt of influenza vaccination.

Aim 3 will measure the effect of adding mailed or text message reminder/recall for autodialer failures vs. autodialer-alone reminder/recall on influenza vaccination rates using a 2-arm randomized controlled trial.

Aim 4 (dissemination aim) will develop a toolkit for state IIS-based influenza vaccine reminder/recall for seasonal and pandemic influenza, and work with key stakeholders on a sustainability plan.

By the end of the study, the investigators will have a feasible and cost-effective model to raise child seasonal or possibly pandemic influenza vaccination rates to prevent influenza. The investigators will disseminate the IIS model to all states.

ELIGIBILITY:
Inclusion Criteria:

* A record in the New York State Immunization Information System
* In need of at least one influenza vaccination at time of study
* Affiliated with a participating practice

Exclusion Criteria:

* Up to date on influenza vaccine

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100000 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects receiving influenza vaccine | 6 months
  The primary outcome is receipt of influenza vaccine by children receiving zero notices compared to those receiving 1,2, or 3 notices.

SECONDARY OUTCOMES:
Number of subjects receiving influenza vaccine based on demographic subgroups | 6 months
  This outcome will categorize the number of influenza vaccines administered by subgroups, e.g. Urban/rural, Pediatrics/Family Practice, and age from 6 months-1.9 years, 2-10.9 years and 11-17.9 years.
Number of subjects <9 years of age that will receive an additional vaccine | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kempe A, Saville A, Dickinson LM, Eisert S, Reynolds J, Herrero D, Beaty B, Albright K, Dibert E, Koehler V, Lockhart S, Calonge N. Population-based versus practice-based recall for childhood immunizations: a randomized controlled comparative effectiveness trial. Am J Public Health. 2013 Jun;103(6):1116-23. doi: 10.2105/AJPH.2012.301035. Epub 2012 Dec 13. PMID 23237154
- [Background] Kempe A, Saville AW, Dickinson LM, Beaty B, Eisert S, Gurfinkel D, Brewer S, Shull H, Herrero D, Herlihy R. Collaborative centralized reminder/recall notification to increase immunization rates among young children: a comparative effectiveness trial. JAMA Pediatr. 2015 Apr;169(4):365-73. doi: 10.1001/jamapediatrics.2014.3670. PMID 25706340
- [Derived] Kempe A, Saville AW, Albertin C, Helmkamp L, Zhou X, Vangela S, Dickinson LM, Tseng CH, Campbell JD, Whittington M, Gurfinkel D, Roth H, Hoefer D, Szilagyi P. Centralized Reminder/Recall to Increase Influenza Vaccination Rates: A Two-State Pragmatic Randomized Trial. Acad Pediatr. 2020 Apr;20(3):374-383. doi: 10.1016/j.acap.2019.10.015. Epub 2019 Nov 5. PMID 31698085